CLINICAL TRIAL: NCT04405414
Title: Observational Study of Cannabidiol Use in Patients Consulting in Addictology and/ or Algology Departments
Brief Title: EffectS of CAnnabidiol in Patients: Evaluation
Acronym: ESCAPE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0405
Record Dates: First submitted 2020-05-15; First posted 2020-05-28 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Substance-Related Disorders
Keywords: Cannabidiol; prevalence; epidemiology; pain; substance-related disorders
MeSH Terms: conditions — Substance-Related Disorders; Pain | interventions — Metabolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Form — Data regarding the use of CBD will be collected: the form, the route of administration, the effects sought and felt, the method of obtaining, the impact on other drugs and/or substances use and the drug liking of CBD

SUMMARY:
Since its recent marketizing in France, the cannabidiol (CBD), a major component of cannabis, is used in many over-the-counter products in France. Some painful patients or patients suffering from addiction seem to use the CBD in search of therapeutic effects. Yet, there are no data available for patients in algology and addictology, particularly with regard to the prevalence of the use of CBD, the effects sought and felt. Faced with the emergence of the use of a substance with a therapeutic purpose but outside a medical framework and without monitoring of adverse effects, it becomes essential to characterize the use of CBD. The main objective of the study is therefore to assess the prevalence of CBD users in algology and addictology departments. Secondary objectives are to characterize the use of CBD as well as the users of CBD, and to evaluate the impact of the use of CBD on other psychoactive substances use or current drug treatments and the drug liking of CBD.

DETAILED DESCRIPTION:
Physicians from algology and addictology departments will propose the study to all patients who meet the inclusion criteria during a medical consultation (in hospitalization or ambulatory care). If the patient agrees to participate, the non-opposition will be collected and the physician will complete a short form with sociodemographic data, medical history and contact details of the patient.

The form will be transmitted securely to the research staff that will perform a unique research evaluation face to face (when the patient is still hospitalized and available) or by phone (when the patient is not available during hospitalization or no longer hospitalized or in case of ambulatory care). The research evaluation includes data about the frequency and the duration of the use of all substances (CBD included) in the last 12 months and the frequency of current drug treatments. For patients with CBD use in the last 12 months, additional data regarding the use of CBD will be collected: the form, the route of administration, the effects sought and felt, the method of obtaining, the impact on other drugs and/or substances use and the drug liking of CBD.

A descriptive analysis will be carried out. The CBD user group and the CBD non-user group will be compared on all the variables collected. A multivariate analysis will be carried out in order to identify factors associated to CBD use in algology and addictology patients.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Patients for whom hospital specialists in algology or addictology have been requested (for hospitalized or ambulatory cares) during the inclusion period.
* Giving oral non opposition to participate.

Exclusion Criteria:

* Adults under guardianship or curator
* Patients unable to respond to the research evaluation (cerebral function disorder, difficulty to understand, read or write French language).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians from algology and addictology departments will propose the study to all patients who meet the inclusion criteria during a medical consultation (in hospitalization or ambulatory care)
Sampling Method: Non-Probability Sample
Enrollment: 746 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of CBD users | through study completion, an average of 2 year
  For all patients included in the study, the use of CBD during the last 12 months (yes or no) will be collected.

SECONDARY OUTCOMES:
Characterization of the use of CBD | through study completion, an average of 2 year
  Prevalence of form, all effects sought and felt, method of obtaining and route of administration of CBD, frequency and duration of the use.
Characterization of CBD users | through study completion, an average of 2 year
  Prevalence of CBD users (use of CBD in the last 12 months) according to patients' characteristics: age categories, sex, employment status, medical history, other psychoactive substances use, current drug treatments.
Impact of the use of CBD | through study completion, an average of 2 year
  Proportion of CBD users who stopped, decreased, increased or initiated drug treatments in relation to the CBD use.
CBD drug-liking | through study completion, an average of 2 year
  Mean on Visual Analog Scale (VAS) on drug liking for CBD and frequency of substances or drug treatments that would be taken as alternatives in the absence of CBD

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France